CLINICAL TRIAL: NCT05340387
Title: Comparison of Balance Resistance Aerobic Cognitive Exercises (BRACE) and Otago's Exercises on Fall Risk Among Elderly Population
Brief Title: Effects of BRACE Protocol on Fall Risk Among Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ghulam Qadir
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Fall Patients
Keywords: BRACE Protocol; Otago's Protocol; Fall Risk; Elderly Population

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Resistance Aerobic Cognitive Exercises (BRACE) (Experimental): BRACE include combination of exercises including, Balance, Resistance, Aerobic, Cognition Exercises.
  Interventions: Other: Balance Resistance Aerobic Cognitive exercises (BRACE)
- Otago's Exercises (Active Comparator): Otago's protocol is combination of warm up, strengthening, balance and flexibility exercises.
  Interventions: Other: Otago's Protocol

INTERVENTIONS:
Other: Balance Resistance Aerobic Cognitive exercises (BRACE) — Study will be conducted after the approval of Ethical review board. The BRACE exercise training would be perform in 4 times a week for 12 weeks, lasting approximately 40-50 minutes each time. Week 1-3 : Balance: Romberg, tandom standing, single leg stance Resistance: chair rise Aerobic exercises: 6mint walk Cognitive: count reverse from 50 Week 4-6: Balance: Sit to stand, functional reach, Tug Test Resistance: stair climbing Aerobic Exercises: Marching in space Cognitive: Remember 5 words, spell backward, remember 5 animals Week 7-9: Balance: Perturbation, throwing a ball, kicking a ball Resistance: Floor transfer, squatting Aerobic Exercises: Cycling Cognitive: Count even number from 1-50, calculation, addition, subtraction, multiplication division Week 10-12: Balance: Combination of All Resistance: Combination of All Aerobic Exercises: 6 minutes' walk test, marching steps, cycling Cognitive: Combination of all
  Arms: Balance Resistance Aerobic Cognitive Exercises (BRACE)
Other: Otago's Protocol — Study will be conducted after the approval of Ethical review board. The Otago's exercise training would be perform in 4 times a week for 12 weeks, lasting approximately 40-50 minutes each time. WEEK 1-3: Warm up: March, head movement, neck movement, back extension, trunk movement, ankle movements Strength: Front knee strengthening, Back knee strengthening, Side hip strengthening, Calf raises, Toe raises (10 repetitions each) Balance: Knee bends, Backwards walking, Walking and turning around, Sideways walking, Tandem stance (heel toe stand), Tandem walk (heel toe walk), One leg stand, Heel walking, Toe walk, Heel toe walking backwards, Sit to stand, Stair walking. (10 repetitions each) Flexibility: calf stretch, back of thigh stretch Hold for 10 to 15 seconds and repeat on other leg.
  Walk: 5 or 10 minutes' walk
  This protocol will be followed for 12 weeks with increased repetitions after every 3 week.
  Arms: Otago's Exercises

SUMMARY:
The objective of this study is to compare the effects of Balance Resistance Aerobic Cognitive Exercises (BRACE) and Otago's exercises on fall risk among elderly population. And to determine the effects of BRACE and Otago's exercise on static and Dynamic balance in elderly population. the study will be randomized control trial including experimental and control group with estimated 17 individual in each group. Balance resistance aerobic resistance exercises will be performed by experimental group and Otago's protocol will be performed by control group.

DETAILED DESCRIPTION:
Balance control is the foundation of a person's ability to move and function independently. However, balance control declines with age, and impaired balance is a major risk factor for falls among older adults. Training balance during dual-task conditions appears to be necessary to improve balance control under situations with divided attention.

Balance training program for older adults, including dual- and multi-task exercises, was designed and developed based on well-established principles of exercise and on the knowledge that balance control relies on the interaction of several physiological systems, as well as interaction with environmental factors and the performed task.

Many studies reported that prevention of fall is possible by adopting a healthy lifestyle, environmental modification, exercise and education. Exercise plays a very important role in fall prevention e.g exercise and tai chi training target balance, flexibility and strength can reduce fall and harm related to fall. Although it does not show a marked difference enjoyable exercise program training is beneficial to achieve healthy outcomes.

A new tool has been designed for fall risk reduction and to mobility in elderly is BRACE (Balance, Resistance, Aerobic, Cognition Exercises). Limited work was done on BRACE protocol so in this study we will do further work on this innovative protocol. The aim of our study is to compare the effects of Balance Resistance Aerobic Cognitive Exercises (BRACE) and Otago's exercises on mobility and fall risk reduction in the elderly

ELIGIBILITY:
Inclusion Criteria:

* berg and balance 0-39

MOCA score not less than 22

Exclusion Criteria:

* • Severe cognitive impairment that prevented them from understanding instructions.

  * Serious musculoskeletal, neurological and visual impairment that might affect measurement.
  * Involvement in other exercise programs.
  * Patients have vertebrobasilar insufficiency
  * Atlanto-axial instability
  * Osteoporosis
  * Rheumatoid arthritis

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Berg And Balance scale | 12 weeks
  changes from the baseline, Berg balance scale (BBS) is used for assessment of balance and fall risk, Higher scores on the BBS indicate greater independence and better ability to balance. In contrast, lower scores indicate a greater fall risk Items DESCRIPTION SCORE (0-4) Sitting to standing, Standing unsupported, Sitting unsupported, Standing to sitting, Transfers , Standing with eyes closed , Standing with feet together, Reaching forward with outstretched arm, Retrieving object from floor, Turning to look behind, Turning 360 degrees, Placing alternate foot on stool, Standing with one foot in front, Standing on one foot, TOTAL __/56
Time Up And Go | 12 week
  changes from the baseline, Timed up and go test is used for the assessment of falls risk among the elderly population. The Timed "Up and Go" (TUG) Test measures, in seconds, the time is taken by an individual to stand up from a standard armchair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down. Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more. Clinical guide: <10 seconds = normal <20 seconds = good mobility, can go out alone, mobile without a gait aid <30 seconds = problems, cannot go outside alone, requires a gait aid A score of more than or equal to 14 seconds has been shown to indicate a high risk of falls.
MOCA | 12 weeks
  The Montreal Cognitive Assessment (MOCA) is a cognitive screening instrument developed to detect mild cognitive impairment (MCI). It is a simple 10 min paper and pencil test that assesses multiple cognitive domains including memory, language, executive functions, visuo-patial skills, calculation, abstraction, attention, concentration, and orientation.
  Scores on the MoCA range from zero to 30. A score of 26 and higher is considered normal.
  In the initial study data, normal controls had an average score of 27.4. People with mild cognitive impairment (MCI) scored an average of 22.1. People with Alzheimer's disease had an average score of 16.2.
Gait dynamic index | 12 weeks
  The DGI tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions.
  It includes eight items, walking on level surfaces, changing speeds, head turns in horizontal and vertical directions, walking and turning 180 degrees to stop, stepping over and around obstacles, and stair ascent and descent.
  Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment. The best possible score on the DGI is a 24.
Activity specific balance scale | 12 weeks
  Activities-specific balance confidence (ABC) scale is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness. It's a 16-item questionnaire where patients' rate their confidence while doing activities. Scoring from 0-100 (0 is no confidence and 100 is full confidence).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute of rehabilitation, Mānsehra, Khyber Pakhtunkhuwa, Pakistan

IPD SHARING:
Plan to Share IPD: No